CLINICAL TRIAL: NCT00317850
Title: Gabapentin for the Relief of Idiopathic Subjective Tinnitus
Brief Title: Gabapentin for the Treatment of Tinnitus
Status: Terminated | Phase: Phase 2 / Phase 3 | Type: Interventional
Sponsor: Washington University School of Medicine (Other)
Collaborators: National Institute on Deafness and Other Communication Disorders (NIDCD) (NIH)
Responsible Party: Principal Investigator, Jay F. Piccirillo, MD, Professor of Otolaryngology, Director of Clinical Outcomes Research Office, Washington University School of Medicine
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Treatment
Other Study IDs: R01DC006253-01 (NIH); R01DC006253 (NIH)
Record Dates: First submitted 2006-04-21; First posted 2006-04-25 (Estimated); Last update posted 2012-03-02 (Estimated); Status verified 2012-02

CONDITIONS: Tinnitus
MeSH Terms: conditions — Tinnitus | interventions — Gabapentin

INTERVENTIONS:
Drug: Gabapentin (Neurontin)

SUMMARY:
The specific aim of the Gabapentin for the Relief of Idiopathic Subjective Tinnitus Trial is to assess the therapeutic benefit of Gabapentin (Neurontin®) for subjective idiopathic troublesome tinnitus. We employed a double-blind placebo-controlled randomized clinical trial design to assess the efficacy of Gabapentin. Adults, between the ages of 18 and 70 with idiopathic, subjective, troublesome, unilateral or bilateral, non-pulsatile tinnitus of 6 month's duration or greater and score of 38 or greater on the Tinnitus Handicap Inventory were enrolled.

ELIGIBILITY:
Inclusion Criteria:

* Adults, between the ages of 18 and 70
* Idiopathic, subjective, troublesome, unilateral or bilateral, non-pulsatile tinnitus (ICD-9 --388.31) of 6 month's duration or greater
* Tinnitus handicap score of 38 or greater on the Tinnitus Handicap Inventory.

Exclusion Criteria:

* The symptoms of tinnitus can be affected by the concomitant use of tricyclic antidepressants, carbamazepine, phenytoin, valproate sodium, or benzodiazepines. Patients who have used these drugs within 30 days of screening will not be enrolled.
* Impaired renal function as determined from serum creatinine levels, using the following formulas35: adult male Ccr = (140 -age) X weight in kilograms/(72 X serum creatinine in milligrams per deciliter); and adult female Ccr = [(140 - age) X weight in kilograms/(72 X serum creatinine in milligrams per deciliter)] X 0.85,whereCcr indicates creatinine clearance.
* Patients with tinnitus related to cochlear implantation, retrocochlear lesion, or other known anatomic/structural lesions of the ear and temporal bone
* Patients with any serious or unstable medical or psychiatric condition.
* Patients whose ability to give informed consent is in question.

Ages: 18 Years to 70 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 160
Dates: Start 2004-04; Study Completion 2006-02

PRIMARY OUTCOMES:
Tinnitus Handicap Inventory Score from Baseline to Week 8

SECONDARY OUTCOMES:
Beck Depression Inventory Score from Baseline to Week 8
Brief Symptom Inventory Score from Baseline to Week 8
Epworth Sleepiness Scale Score from Baseline to Week 8

CONTACTS AND LOCATIONS:
Overall Officials: Jay F Piccirillo, MD, Principal Investigator — Washington University School of Medicine

REFERENCES:
- [Derived] Piccirillo JF, Finnell J, Vlahiotis A, Chole RA, Spitznagel E Jr. Relief of idiopathic subjective tinnitus: is gabapentin effective? Arch Otolaryngol Head Neck Surg. 2007 Apr;133(4):390-7. doi: 10.1001/archotol.133.4.390. PMID 17438255